CLINICAL TRIAL: NCT05623540
Title: Postoperative Use of Bisphosphonates Reduces Adverse Outcome After Primary Total Joint Arthroplasty: A Nationwide Population-based Cohort Study
Brief Title: Bisphosphonates Use After Total Joint Arthroplasty
Status: Completed | Type: Observational
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Jen-Ta Shih, Lecturer, department of Orthopedics, school of Medicine, National Defense Medical Center, Taiwan
Other Study IDs: TSGH-D-110103
Record Dates: First submitted 2022-11-13; First posted 2022-11-21 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Diphosphonates
Keywords: Bisphosphonates; Total joint arthroplasty; Revision surgery; Periprosthetic fracture
MeSH Terms: conditions — Periprosthetic Fractures | interventions — Diphosphonates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bisphosphonates users: Patients who underwent primary total joint arthroplasty with bisphosphonates use
  Interventions: Drug: Bisphosphonates, Combinations
- bisphosphonates nonusers: Patients who underwent primary total joint arthroplasty without bisphosphonates use
  Interventions: Drug: Bisphosphonates, Combinations

INTERVENTIONS:
Drug: Bisphosphonates, Combinations

SUMMARY:
Background Bisphosphonates has been associated with a decreased risk of revision total joint replacements because of its effects on decreased periprosthetic bone loss and prosthetic migration. However, the results in the early literature are inconsistent and the influence of bisphosphonates on associated complications and subsequent total joint arthroplasty (TJA) remains unknown. This study is to investigate the association between the use of bisphosphonates and risk of adverse outcomes after primary TJA.

Materials and Methods This matched cohort study utilized National Health Insurance Research Database in Taiwan to identify patients who underwent primary TJA over a 15-year period (January 2000- December 2015 inclusive). Study participants were further categorized into two groups: bisphosphonates users and nonusers, using propensity score matching. The Kaplan-Meier curve analysis and adjusted hazard ratios (aHR) of revision surgery, adverse outcomes of primary surgery and undergoing subsequent TJA were calculated using Cox regression analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent primary total joint arthroplasty during the study period (January 1, 2000 to December 31, 2015).

Exclusion Criteria:

1. Patients with total joint arthroplasty before the index date,
2. Patients with existing pathologic fracture, nonunion of fracture and partial joint replacement,
3. Patients who were lost to follow-up
4. Patients < 40 years old

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) was used to identify diagnoses and related procedures. The target cohort in NHIRD were those who underwent primary total joint arthroplasty during the study period (January 1, 2000 to December 31, 2015).
Sampling Method: Non-Probability Sample
Enrollment: 27405 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
revision rate of joint arthroplasty | a 15-year period (January 2000- December 2015 inclusive)
  revision rate of joint arthroplasty after primary surgery

SECONDARY OUTCOMES:
The rate of secondary total joint arthroplasty | a 15-year period (January 2000- December 2015 inclusive)
  The rate of secondary total joint arthroplasty
The rate of periprosthetic joint infection | a 15-year period (January 2000- December 2015 inclusive)
  The rate of periprosthetic joint infection
The rate of periprosthetic fracture | a 15-year period (January 2000- December 2015 inclusive)
  The rate of periprosthetic fracture
Mortality rate | a 15-year period (January 2000- December 2015 inclusive)
  Mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no plans to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Shih JT, Tan TL, Shen PH, Yeh TT, Wu CC, Pan RY, Chien WC, Chung CH, Wang SH. Postoperative Bisphosphonates Use is Associated with Reduced Adverse Outcomes After Primary Total Joint Arthroplasty of Hip and Knee: A Nationwide Population-Based Cohort Study. Calcif Tissue Int. 2024 May;114(5):451-460. doi: 10.1007/s00223-024-01192-6. Epub 2024 Mar 16. PMID 38492035